CLINICAL TRIAL: NCT05153122
Title: A Feasibility Study of Evaluation of SenseGuard, Non-Invasive Wearable Device, in Assessing Respiratory Condition Change of Patients With Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: A Feasibility Study of Wearable Device in Assessing Respiratory Condition Change of Patients With Exacerbation of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NanoVation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIV-19-07-029227
Record Dates: First submitted 2021-11-04; First posted 2021-12-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational SenseGuard Device (Experimental): Patients undergo SG monitoring at least twice daily before and after receiving treatment.
  Interventions: Device: SenseGuard

INTERVENTIONS:
Device: SenseGuard — SG is a wireless, wearable medical device, which includes nano-based sensors. It can seamlessly measure patient's tidal breathing during daily activities. SG extracts series of critical respiratory parameters, including; Respiration Rate (RR), Inhalation and Exhalation duration and ratio (I/E), as well as novel biomarkers. SG parameters are applicable to evaluate COPD patients' condition, or for monitoring patients with other respiratory conditions.
  SG components are:
  RSM (Respiratory Sensing Module): non-invasive module with sensors that can detect the exhaled humidity and condensation. The RSM is a non-sterile, disposable, single patient use.
  ECU (Electronic Control Unit): a re-usable, wireless data acquisition and transmission unit. The ECU is connected to the RSM during the measurement and transmits the data via Bluetooth to the SG software.
  SenseGuard™ Software: for data management, acquisition, processing, logging and presentation of the digital respiratory signals.

SUMMARY:
The study will include daily SenseGuard measurement of patients hospitalized with exacerbations of COPD. from admission to discharge. In parallel clinical evaluation of patient's respiratory condition was done daily by routine tests and questionnaires.

DETAILED DESCRIPTION:
A study for evaluating the feasibility of SenseGuard in assessing the respiratory condition change of hospitalized patients with exacerbation of COPD, by monitoring respiratory parameters. The study duration for each patient will start at the time of enrollment until the patient is released, or until the optional post-discharge follow-up visit.

The study will include at least one visit per day: The visit and measurement with SenseGuard will start prior to the first medical exacerbation treatment effect-onset given on each study day (by inhalation or IV). The measurement with SenseGuard will be done before and after treatment.

At the investigator discretion, additional two similar visits could be performed on the same study day, with or without the admission of the medical exacerbation treatment.

During the study, both the investigator and the patients will be asked to fill questionnaires to assess the patient's condition Additionally, measurements that are performed and collected as a standard practice or at the request of the medical personnel as part of patient's treatment course shall be documented and used as a reference for the study device assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Primary or secondary diagnosis of AECOPD (Acute Exacerbation of Chronic Obstructive Pulmonary Disease) in patients with GOLD 1-4/A-D
2. WHO performance status ≤ 3
3. Provision of signed and dated informed consent form.
4. Male or female, aged ≥18.
5. Ability and stated willingness to adhere to the study regimen and availability for the duration of the study.

Exclusion Criteria:

3. Inability to provide informed consent including patients still impacted by the use of narcotics as part of emergency care.

4. Intubated patients or patients undergoing a BIPAP/CPAP/NHF treatment and are medically not able to suspend the treatment for the required duration of the visits or expected intolerance of the sensor in their face due to severe respiratory distress.

5. Presence of implanted electronic device intended to regulate cardiac activity (e.g., pacemaker or cardioverter/defibrillator).

6. Pregnancy or lactation. 7. Known allergic reactions to materials used in the components of the SenseGuard™ system, i.e. polyethylene or silicon, or gold, nickel, copper or alloys containing any of the above.

8. Participation in another study that is related to treatment of the respiratory condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of SenseGuard respiratory parameter - Respiratory Rate, in the measurement of clinical change in COPD patients hospitalized with AECOPD | 24 months
  SenseGuard respiratory parameters (Respiratory Rate in BPM ) can be used to assess the changes in respiratory condition of 80% of exacerbated COPD patient, as defined by physician's assessment, patient's self-assessment and/or as measured by current conventional methods.
Evaluation of SenseGuard respiratory parameter - Inhalation to Exhalation ratio, in the measurement of clinical change in COPD patients hospitalized with AECOPD | 24 months
  SenseGuard respiratory parameters (Inhalation and Exhalation time and ratio) can be used to assess the changes in respiratory condition of 80% of exacerbated COPD patient, as defined by physician's assessment, patient's self-assessment and/or as measured by current conventional methods.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Eisenmann, Dr., Principal Investigator — Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Innere Medizin I
Locations (2):
- Universitätsklinikum Halle (Saale) Universitätsklinik und Poliklinik für Innere Medizin I, Halle, Germany
- Galilee Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Undecided